CLINICAL TRIAL: NCT04209283
Title: Using a Visuospatial Interference Intervention to Reduce Intrusive Memories Among Trauma Exposed Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Responsible Party: Principal Investigator, Andri Steinþór Björnsson, Professor, University of Iceland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UI-2019-VIRM
Record Dates: First submitted 2019-12-06; First posted 2019-12-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Trauma
Keywords: Intrusive memories
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma exposed women (Experimental): No Intervention: Baseline phase ('A'):
  Measurements collected in a daily diary four times a day (morning, afternoon, evening and night) over one week for the primary outcome (occurrence of intrusive memories of trauma). Individual baseline phases will be used as control periods.
  Experimental: Intervention phase ('B'):
  A one-session intervention with a researcher including a simple cognitive task (a memory cue and 25 minutes of Tetris game-play with mental rotation) followed by instructions to engage in the task self-guided over the subsequent week. Measurements collected in a daily diary four times a day following the intervention for the primary outcome (occurrence of intrusive memories of trauma).
  Intervention: Behavioral: Brief cognitive intervention
  Interventions: Behavioral: Visuospatial interference

INTERVENTIONS:
Behavioral: Visuospatial interference — Behavioral: Brief cognitive intervention. A one-session intervention with a researcher including a simple cognitive task (a memory cue and 25 minutes of Tetris game play with mental rotation) with instructions to engage in the task self-guided in the subsequent weeks.

SUMMARY:
This research study is designed to investigate the use of a simple cognitive task (a memory cue followed by playing the computer game "Tetris") for decreasing the number of intrusive memories of trauma among trauma-exposed women in Iceland. This is a single case series using a within subject multiple baseline AB design. Participants will aim to complete a no-intervention phase ('A': baseline phase) of one week followed by a one-week intervention phase ('B'), including a one-session intervention with a researcher comprising the simple cognitive task, followed by instructions to continue using the technique self-guided in subsequent weeks. Participants will be asked to monitor the occurrence of intrusive memories of trauma in a daily diary. It is predicted that participants will report fewer intrusive memories during the intervention phase than during the preceding baseline phase and that the frequency of targeted intrusive memories is going to decrease relative to non-targeted intrusive memories. Furthermore, we will explore whether having fewer intrusive memories has an impact on function and/or PTSD, depressive or anxiety symptoms.

DETAILED DESCRIPTION:
Participants will attend 3-8 sessions with the researcher. In session one, the intrusive memories will be logged for monitoring their frequency in a daily diary for the following weeks. Baseline assessment questionnaires will also administered. In the second session, a memory will be selected and targeted with the intervention (memory reminder followed by 25 min gameplay with mental rotation) followed by monitoring the frequency of both the targeted and non-targeted intrusive memories. Participants will also complete self-rated questions concerning the impact of their intrusive memories. The intervention session will be repeated for other intrusive memories (maximum 6 intervention sessions). In the last intervention session, participants will be asked to complete questionnaires and self-rated questions assessing the impact of their intrusive memories. Participants will be asked to complete measures at 1 month follow-up and at 3 month follow-up. In the 1 month follow-up, participants complete questionnaires and monitor the frequency of intrusive memories for one week in the daily diary.

The previous version of the CTR incorrectly stated that at the 3 month time point the measure of intrusions will be: 'Questions about the frequency of intrusive memories for the past day/week (for each intrusive memory, to be tallied to arrive at a mean frequency for the memories for the previous day and for the week)'. We changed this measure at the study start to using the same diary as we used for the earlier time points (i.e., daily diary with the same level of detail as the ones used at e.g. at 1 month), but failed to update this in the CTR. The measure has been updated retrospectively in the CTR for this timepoint, and should be interpreted with caution accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Having experienced at least one criterion A trauma according to the DSM-5
* Having at least one intrusive memory that occurs at least three times per week in the past four weeks
* Being able to attend 3-8 sessions with researcher
* Being willing to monitor intrusive memories in daily life
* Having access to a smartphone
* Being able to speak Icelandic and read study materials in Icelandic

Exclusion Criteria:

* Current psychotic disorder (determined by the psychotic module on the Mini International Neuropsychiatric Interview (MINI)).
* Current manic episode (determined by the bipolar module on the Mini International Neuropsychiatric Interview (MINI)).
* Being acutely suicidal (according to the module assessing suicidality on the Mini International Neuropsychiatric Interview (MINI)).

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Change in the number of intrusive memories of trauma | Baseline week 1; Intervention week 1-6 and 1 month follow-up
  Number of intrusive memories of traumatic event recorded by participants in a diary daily (morning, afternoon, evening and night) for one week during the baseline phase and each week during the intervention phase (week 1-6) and during one week at one month follow-up.
Change in the number of intrusive memories of trauma from baseline to 3 month follow up | Baseline week 1; 3 month follow-up
  Number of intrusive memories of traumatic event recorded by participants in a diary daily (morning, afternoon, evening and night) per week during the baseline phase and during one week at three month follow-up.
  Note that the way this outcome was measured had been specified incorrectly in the previous versions of this CTR (as using questions about frequency) and was therefore updated retrospectively after the end of data collection to the same diary as the previous time points.

SECONDARY OUTCOMES:
Self-guided intervention adherence - usage of the gameplay intervention in daily life | Intervention week 2-6
  How often did you manage to play Tetris after you experienced an intrusive memory? (11-point scale; 0 = not at all; 10 = every time).
Feasibility and acceptability ratings for using a smartphone game-play intervention | Post intervention up to week 7
  Feasibility and Acceptability of the intervention assessed with two self-rated items, "Would you recommend playing Tetris to a friend?" and "Do you consider gameplay to be an acceptable way to reduce the daily frequency of intrusive memories?". Scores could range from 0 - 10 with higher scores indicating greater acceptability/feasibility.
Feasibility and acceptability - open ended questions | Post intervention up to week 7
  Two open-ended questions: 1. "How did you feel about playing Tetris after you had an intrusive memory?" 2. "Did you find the intervention helpful? If yes, how?"
Impact of intrusive memories on concentration, sleep and stress - ratings | Baseline week 1; Post intervention up to week 7; 1 month follow-up and 3 month follow-up
  Six self-rated items to assess the impact of intrusive memories on concentration, sleep, and stress in the past week. 2 items assessing concentration difficulties in general and due to intrusive memories (11-point scale; high scores indicating more difficulties). 2 items assessing sleep disturbances due to intrusive memories (11-point scale; higher scores indicating more sleep disturbance); and 1 item assessing to what degree intrusive memories affected stress levels (0 = not at all; 10 = affected very much).
Rating of how long intrusive memories disrupted concentration on average | Baseline week 1; Post intervention up to week 7; 1 month follow-up and 3 month follow-up
  1 item assessing for how long intrusive memories disrupted concentration on average (<1 minute - > 60 minutes)
General impact of intrusive memories - ratings | Baseline week 1; Intervention week 1-6; 1 month follow-up and 3 month follow-up
  Two items both rated on an 11-point scale: 1. "During the last week, how distressing were your intrusive memories (0 = not at all; 10 = very distressing). 2. During the last week, how vivid were your intrusive memories (0 = not at all; 10= very vivid)
Intrusion diary adherence | Baseline phase week 1; Intervention week 1-6 and 1 month follow-up
  Adherence to the intrusion diary assessed with 1 item: "How accurately did you fill out the diary?" (0= not at all; 10 = very accurately)
The Posttraumatic Stress Disorder Checklist 5 (PCL-5) | Baseline week 1; Post intervention up to week 7 and 1 month follow-up
  The PCL-5 is a short 20-item self-report scale used to assess the severity of PTSD symptoms corresponding to the DSM-5 criteria for PTSD. Symptoms are rated from 0-4. Higher scores indicate greater severity.
The Patient Health Questionnaire-9 (PHQ-9) | Baseline week 1; Post intervention up to week 7 and 1 month follow-up
  The PHQ-9 is a 9-item self-report measure of depression symptoms and the severity of those symptoms. Each item can be scored from 0 (i.e., not at all) to 3 (i.e., nearly every day).
The Generalized Anxiety Disorder-7 scale (GAD-7) | Baseline week 1; Post intervention up to week 7 and 1 month follow-up
  The GAD-7 is a brief self-report questionnaire designed as a screening tool for symptoms of general anxiety disorder and their severity. Each item can be scored from 0 (i.e., not at all) to 3 (i.e., nearly every day).
The Sheehan Disability Scale (SDS) | Baseline week 1; Post intervention up to week 7 and 1 month follow-up
  The SDS is a self-report questionnaire which is designed to assess functional impairment across three domains: (1) Work/school, (2) social, and (3) family life. These domains are measured on an 11-point scale which ranges from 0 (i.e., not at all) to 10 (i.e., extremely). The scale will be adjusted to assess impairment associated with intrusive memories.
Impact of intrusive memories on functioning | Baseline week 1; Post intervention up to week 7, 1 month follow-up and 3 month follow-up
  Two questions assessing the impact intrusive memories have on functioning in daily life. One question is open-ended: "How have the intrusive memories affected your ability to function in your daily life in the past week?" and one question is self-rated: "Have the intrusive memories affected your ability to function in your daily life?" (11-point scale, higher score indicate greater impact on functioning.)

CONTACTS AND LOCATIONS:
Overall Officials: Andri Björnsson, PhD, Principal Investigator — University of Iceland Sæmundargata 12 101 Reykjavík, Iceland
Locations (1):
- University of Iceland, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No